CLINICAL TRIAL: NCT01883102
Title: The Effect of Ablation of Epidermal Nerve Fibers Using 0.1% Capsaicin Cream on Spontaneous Cutaneous Burning Pain, Tactile Hyperalgesia, and Thermal Hyperalgesia: A Controlled, Masked Trial With an N of 1
Brief Title: The Effect of Ablation of Epidermal Nerve Fibers Using Capsaicin Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Peter J. Dyck, M.D., MD, Mayo Clinic
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: 13-002235
Record Dates: First submitted 2013-06-06; First posted 2013-06-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capsaicin 0.1% (Experimental): Capsaicin cream 0.1% will be applied to site A or B on the subject's abdomen daily for 7 days.
  Interventions: Drug: Capsaicin 0.1%
- Placebo/cream without 0.1% capsaicin (Placebo Comparator): The placebo cream will be applied to site A or B on the subject's abdomen daily for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Capsaicin 0.1% — Cream will be cleansed from sites A and B with soap and water each morning before reapplying.
  Other Names: Capzacin
  Arms: Capsaicin 0.1%
Drug: Placebo — Cream will be cleansed from sites A and B with soap and water each morning before reapplying.
  Arms: Placebo/cream without 0.1% capsaicin

SUMMARY:
This is a study of epidermal (the outer most layer) nerve fibers (ENFs) in the skin of the body; counts of which are used to determine a disease of nerves called "small nerve fiber neuropathy."

Capsaicin is approved by the Food and Drug Administration (FDA) for pain relief. Since 0.1% capsaicin is known to cause ablation (removal) of ENFs, this study will test whether such ablation results in relief of spontaneous pain, touch, or heat-pain.

DETAILED DESCRIPTION:
On the first day, two areas of the skin of the subject's right abdomen will be marked and identified as sites A and B. Each day for one week the subject will be asked to grade her degree of discomfort or pain from 1 to 10 at sites marked A and B every two hours beginning at 8 a.m. and ending at 10 p.m.

Each day except for Saturday and Sunday touch-pressure sensation will be evaluated using monofilaments and heat pain sensation at sites A and B. Also evaluated will be touch pressure pain at each of these sites.

On Thursday of the first week 3 mm punch biopsies of the skin will be obtained from sites A and B and another 3 mm punch biopsy will be obtained on Thursday of the following week from sites A and B.

Following the first biopsy, the experimental creams will be applied to sites A and B. One of the experimental creams contains 0.1% Capsaisin in a bland cream. The second cream contains no Capsaisin. 0.1% Capsaisin is known to destroy the small fibers, especially pain fibers in the skin. Both the investigators applying the cream and the subject will not know which experimental cream contains the Capsaisin. The creams will be applied on Thursday of the first week but only after all testing and skin biopsies have been done. The creams will be left in place except when testing is being done, and they will not be applied after the second set of skin biopsies has been obtained.

The creams will be applied by the investigators and by the subject, care being taken so that the tube marked A is applied to the site marked A, and the tube marked B is applied to the site marked B. Between application to the two sites, investigators and the subject will use different gloves and applicators, carefully washing their hands with soap and water between and after applications.

The subject will be asked not to shower or to immerse herself in water but to use sponge baths, avoiding the tested areas, so that the cream does not move to other areas.

ELIGIBILITY:
Inclusion Criteria:

* pain syndrome
* must be able to be in study for one week

Exclusion Criteria:

- not able to be in study for one week

Min Age: 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Burning pain as measured by a numeric rating scale of 1-10 | 1 week

SECONDARY OUTCOMES:
Tactile hyperalgesia as measured with monofilaments A, B, C, (through I), ranging in providing forces -3, -2, -1 (through +5) In grams | 1 week
  This outcome measure consists of touch pressure testing of tactile hyperalgesia (increased sensitivity to pain) with monofilaments consists of recognizing the lowest level at which the subject can feel the touch of a monofilament hair, and to the point of discomfort or pain.
  The units for tactile hyperalgesia are In grams of touch pressure.
Thermal hyperalgesia as measured by the heat as pain thermode test using CASE IVc | 1 week
  This outcome measure tests heat-pain sensation (the lowest degree of a thermal warming pulse that the subject can perceive as discomfort or pain).
  CASE IVc is a computerized quantitative sensation testing instrument, extensively described. It was originally developed at Mayo Clinic and the Section of Engineering. It is now manufactured by WR Medical Electronics in Maplewood, Minnesota. This instrument provides exponentially increasing pyramidal and trapezoid heat pulses to a maximum of 49 degrees centigrade for 10 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Dyck, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States